CLINICAL TRIAL: NCT04493216
Title: A Phase IIb, Randomized, Partially Blind, Active Controlled, Dose-range Finding Study of GSK3640254 Compared to a Reference Arm of Dolutegravir, Each in Combination With Nucleoside Reverse Transcriptase Inhibitors, in HIV-1 Infected Antiretroviral Treatment-naive Adults
Brief Title: A Dose-Range Finding Clinical Trial Study in Human Immunodeficiency Virus (HIV-1) Infected Treatment-Naive Adults
Acronym: DOMINO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to stop compound development. The decision is not based on any safety or efficacy concerns. It reflects the company strategy for portfolio progression.
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 208379
Record Dates: First submitted 2020-07-10; First posted 2020-07-30 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
Keywords: HIV infection; GSK3640254; Nucleoside Reverse Transcriptase Inhibitor; Dolutegravir; Abacavir (ABC)/Lamivudine (3TC); Emtricitabine (FTC)/tenofovir alafenamide (TAF); Maturation Inhibitor
MeSH Terms: conditions — HIV Infections | interventions — GSK3640254; dolutegravir

STUDY DESIGN:
Intervention Model Description: This is a randomized, multicenter, parallel group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study treatment assignments was not blinded (GSK3640254 versus Dolutegravir control arm). However, the dose level of GSK3640254 in each of the treatment arms containing GSK3640254 was blinded to the research participants and all study personnel during the study. The Sponsor personnel remained blinded until the database lock for the Week 24 analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF (Experimental): Participants with human immunodeficiency virus type 1 (HIV-1), orally received one 100 mg tablet per day of GSK3640254 and two tablets per day of matching placebo in a blinded setting. Open label dual NRTI background therapies were given as one tablet per day of 600 mg abacavir (ABC) / 300 mg lamivudine (3TC) OR 200 mg emtricitabine (FTC) / 25 mg tenofovir alafenamide (TAF) orally.
  Interventions: Drug: GSK3640254; Drug: ABC/3TC; Drug: FTC/TAF; Drug: Placebo
- GSK3640254 150 mg + ABC/3TC or FTC/TAF (Experimental): Participants with HIV-1, orally received 150 mg (one 100 mg tablet + two 25 mg tablets per day) of GSK3640254 in a blinded setting. Open label dual NRTI background therapies were given as one tablet per day combination of 600 mg ABC / 300 mg 3TC OR 200 mg FTC / 25 mg TAF orally.
  Interventions: Drug: GSK3640254; Drug: ABC/3TC; Drug: FTC/TAF
- GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF (Experimental): Participants with HIV-1, orally received two 100 mg tablets (200 mg) per day of GSK3640254 and one tablet per day of matching placebo in a blinded setting. Open label dual NRTI background therapies were given as one tablet per day combination of 600 mg ABC / 300 mg 3TC OR 200 mg FTC / 25 mg TAF orally.
  Interventions: Drug: GSK3640254; Drug: ABC/3TC; Drug: FTC/TAF; Drug: Placebo
- Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF (Active Comparator): Participants with HIV-1, orally received one 50 mg tablet per day of DTG in an open label setting. Open label dual NRTI background therapies were given as one tablet per day combination of 600 mg ABC / 300 mg 3TC OR 200 mg FTC / 25 mg TAF orally.
  Interventions: Drug: ABC/3TC; Drug: FTC/TAF; Drug: Dolutegravir

INTERVENTIONS:
Drug: GSK3640254 — GSK3640254 was available as a 25 mg and 100 mg tablets to be administered via oral route.
  Arms: GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF; GSK3640254 150 mg + ABC/3TC or FTC/TAF; GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF
Drug: ABC/3TC — ABC/3TC was available as abacavir 600 mg/lamivudine 300 mg tablet to be administered via oral route.
Drug: FTC/TAF — FTC/TAF was available as emtricitabine 200 mg/tenofovir alafenamide 25 mg tablet to be administered via oral route.
Drug: Dolutegravir — Dolutegravir was available as a 50 mg tablet to be administered via oral route.
  Arms: Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Drug: Placebo — Placebo matching GSK3640254 was administered in the form of tablets via oral route.
  Arms: GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF; GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF

SUMMARY:
This is a phase 2b, randomized, multicenter, parallel group, partially blind (to GSK3640254 doses [100, 150 and 200 milligrams {mg}]), active controlled clinical trial. It aims to investigate the safety, efficacy and dose-response of GSK3640254 compared to dolutegravir (DTG), each given in combination with 2 Nucleoside Reverse Transcriptase Inhibitors (NRTIs) (abacavir/lamivudine [ABC/3TC] or emtricitabine/tenofovir alafenamide [FTC/TAF]).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age inclusive, at the time of signing the informed consent.
* Treatment-naive, defined as no anti-retrovirals (ARVs) (in combination or monotherapy) received after the diagnosis of HIV-1 infection (for example [e.g.], use of Pre-exposure prophylaxis [PreP] meets inclusion.
* Documented HIV infection and Screening plasma HIV-1 RNA greater than or equal to (>=)1000 c/mL.
* Screening CD4+ T-cell count >=250 cells/mm^3.
* Antiviral susceptibility to the NRTI backbone selected should be demonstrated
* Body weight >=50.0 kilograms (kg) (110 pounds [lbs]) for men and >=45.0 kg (99 lbs) for women and body mass index (BMI) greater than (>)18.5 kg/meter square (m^2).Calculations utilized sex assigned at birth
* Participants who are male at birth and participants who are female at birth.
* Participants who are female at birth: Contraceptive use by participant who are female at birth should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  • A participant who was female at birth was eligible to participate if they were not pregnant or breastfeeding, and one of the following conditions applies:
  * Was a participant of non-childbearing potential (PONCBP)
  * Or was a POCBP and using an acceptable contraceptive method during the study intervention period (at a minimum until after the last dose of study intervention).
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* For participants enrolled in France: a participant was eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion criteria:

* Any evidence of an active Center for Disease Control and Prevention (CDC) Stage 3 disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia.
* Presence of primary HIV-1 infection, evidenced by acute retroviral syndrome (e.g., fever, malaise, fatigue) and/or evidence of recent (within 3 months) documented viremia without antibody production and/or evidence of recent (within 3 months) documented seroconversion.
* Known history of liver cirrhosis with or without viral hepatitis co-infection.
* Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* History of ongoing or clinically relevant hepatitis within the previous 6 months.
* History of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
* Any history of significant underlying psychiatric disorder, in the opinion of the Investigator or ViiV Medical Monitor, including but not limited to schizophrenia, bipolar disorder with or without psychotic symptoms, other psychotic disorders, or schizotypal (personality) disorder or a clinical assessment of suicidality based on the responses on the Columbia-Suicide Severity Rating Scale (eCSSRS).
* Any history of major depressive disorder with or without suicidal features, or anxiety disorders, that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (>6 months) outpatient treatment.
* Any pre-existing physical or other psychiatric condition (including alcohol or drug abuse), which, in the opinion of the Investigator or ViiV Medical Monitor (with or without psychiatric evaluation), could interfere with the participant's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the participant.
* A pre-existing condition, in the opinion of the Investigator or ViiV Medical Monitor, that could interfere with normal gastrointestinal anatomy or motility (e.g., gastroesophageal reflux disease [GERD], gastric ulcers, gastritis, inflammatory bowel disease), hepatic and/or renal function, or with the absorption, metabolism, and/or excretion of the study drugs or render the participant unable to take oral study treatment.
* Myocardial infarction in the past 3 months.
* Familial or personal history of long QT syndrome or sudden cardiac death.
* Medical history, current or historical, of significant cardiac arrhythmias or Electrocardiogram (ECG) findings which, in the opinion of the Investigator or ViiV Medical Monitor, will interfere with the safety of the participant.
* Active Treatment for a viral infection other than HIV-1, such as Hepatitis B, with an agent that is active against HIV-1 (were known to be infected with HIV-1 after treatment for Hepatitis B was completed).
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
* Treatment with any of the following agents within 28 days of Screening: radiation therapy, cytotoxic chemotherapeutic agents, any systemic immune suppressant.
* Participants receiving any protocol-prohibited medication and who are unwilling or unable to switch to an alternate medication.
* Participants who are unwilling to stop any medications as required by the local lab test for Helicobacter (H.) pylori.
* Participants who require concomitant medications known to be associated with a prolonged Corrected QT interval (QTc).
* Exposure to an experimental drug, human blood product, monoclonal antibody, or vaccine (which does not have emergency, conditional or standard market authorization) within 28 days prior to the first dose of study treatment.
* Current enrollment or past participation within the last 30 days before signing of consent in any other clinical study involving an investigational study intervention (including an investigational Coronavirus Disease (COVID) vaccine) or any other type of medical research.
* Any evidence of viral resistance based on the NRTI backbone selected.
* Historical evidence (prior to study screening period) of the presence of resistance- associated mutations gag A364V or A364A/V.
* Creatinine Clearance <50 mL/minute.
* Alanine aminotransferase (ALT) >=3 times upper limit of normal (ULN) or ALT >=2 times ULN and total bilirubin >=1.5 times ULN.
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antibody (anti-HBs) and reflex HBV deoxyribonucleic acid (DNA) as follows:

  1. Participants positive for HBsAg were excluded;
  2. Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA on reflex testing were excluded.
* Positive Hepatitis C antibody test result at Screening and positive on reflex to Hepatitis C RNA.
* Positive test results for H. pylori;
* Known or suspected active COVID-19 infection or contact with an individual with known COVID-19, within 14 days of study enrollment
* Untreated syphilis infection (positive rapid plasma reagin [RPR] at Screening) without documentation of treatment.
* Presence of moderate-to-severe hepatic impairment (Class B or C) as determined by Child-Pugh classification.
* Any acute laboratory abnormality at Screening, which, in the opinion of the investigator or ViiV Medical Monitor, would preclude participation in the study of an investigational compound.
* Urine Drug Screen positive (showing presence of): Amphetamines, Barbiturates, Cocaine, 3,4-Methyl enedioxy methamphetamine (MDMA) or Phencyclidine, or non-prescribed opiates, oxycodone, benzodiazepines, methadone, methamphetamines or tricyclic antidepressants.
* Any clinically relevant Grade 4 laboratory abnormality at Screen, including results for creatine phosphokinase (CPK) and lipid abnormalities that lack a compelling explanation from the Investigator.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 28 days.
* Exposure to more than 4 new investigational drugs or vaccines (exclusive of a severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) potential indication within 12 months prior to the first dosing day;
* Treatment with radiation therapy or cytotoxic chemotherapeutic agents or any systemic immunosuppressive agent within 30 days of study drug administration or anticipated need for such treatment within the study;
* ECG Heart Rate <50 beats per minute (bpm) or >100 bpm, or QT duration corrected for heart rate by Fridericia's formula (QTcF) >450 milliseconds (msec).
* For Portugal only: HIV-2 infection (either determined by prior testing, medical history, or obtained locally during the Screening window).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2023-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (50):
- United States (8):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Berkley, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dallas, Texas
- Argentina (5):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, San Juan
- Canada (2):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (3):
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Tourcoing
- Germany (3):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
- Italy (5):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Milan
- Portugal (3):
  - GSK Investigational Site, Almada
  - GSK Investigational Site, Aveiro
  - GSK Investigational Site, Porto
- Russia (4):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Smolensk
- South Africa (4):
  - GSK Investigational Site, Johannesburg, Gauteng
  - GSK Investigational Site, Wentworth, KwaZulu-Natal
  - GSK Investigational Site, Observatory, Cape Town
  - GSK Investigational Site, Vosloorus Ext 2
- Spain (12):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona, Barcelona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Joshi SR, Cordova E, Mitha E, Castagna A, Ramgopal M, Llibre JM, Potthoff A, Chernova OE, Nunez SA, Man C, Jeffrey JL, Fishman C, Oyee J, Joshi A, Zhang Y, Bainbridge V, Wynne B, Lataillade M. Efficacy and safety of the HIV-1 maturation inhibitor GSK3640254 plus two NRTIs in adults naive to antiretroviral therapy (DOMINO): 24-week results from a randomised phase 2b study. EClinicalMedicine. 2025 Oct 17;89:103567. doi: 10.1016/j.eclinm.2025.103567. eCollection 2025 Nov. PMID 41357330
- [Derived] Spinner CD, Felizarta F, Rizzardini G, Philibert P, Mitha E, Domingo P, Stephan CJ, DeGrosky M, Bainbridge V, Zhan J, Dumitrescu TP, Jeffrey JL, Xu J, Halliday F, Gan J, Johnson M, Gartland M, Joshi SR, Lataillade M. Phase IIa Proof-of-Concept Evaluation of the Antiviral Efficacy, Safety, Tolerability, and Pharmacokinetics of the Next-Generation Maturation Inhibitor GSK3640254. Clin Infect Dis. 2022 Sep 14;75(5):786-794. doi: 10.1093/cid/ciab1065. PMID 34996113

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study assessed efficacy, safety and resistance of GSK3640254 in combination with ABC/3TC or FTC/TAF compared to dolutegravir + ABC/3TC or FTC/TAF in HIV-1 infected, treatment-naïve adults. The study was terminated by the sponsor at Week 48 as the sponsor determined further development of GSK3640254-containing daily oral regimen would not be differentiated enough from existing 2-drug daily oral regimens. Thus, secondary analyses at Week 96 and Week 144 were not evaluated.
Pre-assignment Details: The changes from the planned subsequent analyses were presented as pre-specified in Statistical Analysis Plan. Safety analysis is presented based on the Entire Duration of Treatment Exposure period, which was defined from Day 1 up to end of continued access to treatment post-study termination (Day 922).
Period: Overall Study
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Started | 40 | 43 | 42 | 36
Completed | 0 | 0 | 0 | 0
Not Completed | 40 | 43 | 42 | 36
Not completed — Study terminated by sponsor | 30 | 33 | 28 | 27
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 2
Not completed — Protocol Violation | 1 | 2 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 1
Not completed — Adverse Event | 1 | 4 | 5 | 2
Not completed — Subject reached protocol-defined stopping criteria | 4 | 2 | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF | Total
Number analyzed (Participants) | 40 | 43 | 42 | 36 | 161
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 32.8 (6.20) | 38.1 (12.54) | 33.7 (10.59) | 35.3 (9.85) | 35.0 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 12 | 10 | 38
  Male | 33 | 34 | 30 | 26 | 123
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 1 | 2 | 1 | 0 | 4
  ASIAN | 0 | 2 | 2 | 1 | 5
  BLACK OR AFRICAN AMERICAN | 6 | 8 | 6 | 6 | 26
  WHITE | 32 | 31 | 32 | 29 | 124
  MIXED RACE | 1 | 0 | 0 | 0 | 1
  MISSING | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma HIV-1 Ribonucleic Acid (RNA) Less Than (<)50 Copies Per Milliliter (c/mL) at Week 24
Description: Percentage of participants with plasma HIV-1 RNA <50 c/mL at week 24 was assessed using the Food and Drug Administration (FDA) snapshot algorithm to demonstrate the antiviral activity of GSK3640254 given in combination with either ABC/3TC or FTC/TAF compared to the reference treatment of DTG given in combination with either ABC/3TC or FTC/TAF.
Time Frame: At Week 24
Population: The analysis was performed on the Intent-to-Treat Exposed (ITT-E) population which included all randomized participants who received at least one dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Number analyzed (Participants) | 40 | 43 | 42 | 36
Percentage of participants | 82.5 [68.1 to 91.3] | 90.7 [78.4 to 96.3] | 76.2 [61.5 to 86.5] | 91.7 [78.2 to 97.1]
Statistical Analysis 1: Comparison: GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF vs Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF; Test type: Other; Differences in percentage of participant = -9.2, 95% CI 2-sided [-24.0 to 5.7] — Differences in percentage of participant = Percentage of participant in GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF - Percentage of participant in DTG+ABC/3TC or FTC/TAF
Statistical Analysis 2: Comparison: GSK3640254 150 mg + ABC/3TC or FTC/TAF vs Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF; Test type: Other; Differences in percentage of participant = -1.0, 95% CI 2-sided [-13.5 to 11.6] — Differences in percentage of participant = Percentage of participant in GSK3640254 150 mg+ ABC/3TC or FTC/TAF - Percentage of participant in DTG+ ABC/3TC or FTC/TAF
Statistical Analysis 3: Comparison: GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF vs Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF; Test type: Other; Differences in percentage of participant = -15.5, 95% CI 2-sided [-31.2 to 0.3] — Differences in percentage of participant = Percentage of participant in GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF - Percentage of participant in DTG+ ABC/3TC or FTC/TAF

2. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Week 48
Description: Percentage of participants with plasma HIV-1 RNA <50 c/mL at week 48 was assessed using the FDA snapshot algorithm to demonstrate the antiviral activity of GSK3640254 given in combination with either ABC/3TC or FTC/TAF compared to the reference treatment of DTG given in combination with either ABC/3TC or FTC/TAF.
Time Frame: At Week 48
Population: The analysis was performed on the ITT-E population which included all randomized participants who received at least one dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Number analyzed (Participants) | 40 | 43 | 42 | 36
Percentage of participants | 85.0 [70.9 to 92.9] | 83.7 [70.0 to 91.9] | 76.2 [61.5 to 86.5] | 77.8 [61.9 to 88.3]

3. Secondary Outcome: Absolute Values of HIV-1 RNA at Weeks 24 and 48
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Logarithm to base 10 (log10) values for plasma HIV-1 RNA have been presented. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: The analysis was performed on the ITT-E population which included all randomized participants who received at least one dose of study intervention. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Log 10 copies per milliliter
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Number analyzed (Participants) | 40 | 43 | 42 | 36
Log 10 copies per milliliter
  Baseline (Day 1) | 4.351 (0.5712) | 4.353 (0.6705) | 4.165 (0.6505) | 4.247 (0.6765)
  Week 24: number analyzed (Participants) | 38 | 39 | 33 | 31
  Week 24 | 1.619 (0.1260) | 1.607 (0.0663) | 1.610 (0.0679) | 1.592 (0.0126)
  Week 48: number analyzed (Participants) | 33 | 37 | 31 | 28
  Week 48 | 1.602 (0.0536) | 1.605 (0.0647) | 1.594 (0.0233) | 1.590 (0.0000)

4. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA at Weeks 24 and 48
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. log10 values for plasma HIV-1 RNA have been presented. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Log 10 copies per milliliter
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Number analyzed (Participants) | 40 | 43 | 42 | 36
Log 10 copies per milliliter
  Baseline (Day 1) | 4.351 (0.5712) | 4.353 (0.6705) | 4.165 (0.6505) | 4.247 (0.6765)
  Change from Baseline to Week 24: number analyzed (Participants) | 38 | 39 | 33 | 31
  Change from Baseline to Week 24 | -2.718 (0.5501) | -2.784 (0.6615) | -2.565 (0.6513) | -2.629 (0.6835)
  Change from Baseline to Week 48: number analyzed (Participants) | 33 | 37 | 31 | 28
  Change from Baseline to Week 48 | -2.675 (0.5640) | -2.762 (0.6784) | -2.580 (0.6941) | -2.717 (0.6672)

5. Secondary Outcome: Absolute Values of Cluster of Differentiation 4 Plus (CD4+) Cell Counts at Weeks 24 and 48
Description: Blood samples were collected and CD4+ cell count was assessed using flow cytometry. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Number analyzed (Participants) | 40 | 43 | 42 | 36
Cells per cubic millimeter
  Baseline (Day 1) | 480.3 (171.72) | 509.7 (207.13) | 478.7 (204.04) | 514.1 (240.88)
  Week 24: number analyzed (Participants) | 36 | 37 | 34 | 31
  Week 24 | 717.5 (222.91) | 643.5 (202.27) | 689.8 (316.64) | 724.8 (403.99)
  Week 48: number analyzed (Participants) | 32 | 36 | 30 | 28
  Week 48 | 749.9 (328.28) | 702.6 (258.65) | 747.3 (313.15) | 705.2 (221.18)

6. Secondary Outcome: Change From Baseline in CD4+ Cell Counts at Weeks 24 and 48
Description: Blood samples were collected and CD4+ cell count was assessed using flow cytometry. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Number analyzed (Participants) | 40 | 43 | 42 | 36
Cells per cubic millimeter
  Baseline (Day 1) | 480.3 (171.72) | 509.7 (207.13) | 478.7 (204.04) | 514.1 (240.88)
  Change from Baseline to Week 24: number analyzed (Participants) | 36 | 37 | 34 | 31
  Change from Baseline to Week 24 | 241.3 (191.26) | 129.3 (233.07) | 202.3 (271.98) | 198.5 (285.00)
  Change from Baseline to Week 48: number analyzed (Participants) | 32 | 36 | 30 | 28
  Change from Baseline to Week 48 | 292.4 (264.16) | 189.2 (216.10) | 243.0 (233.24) | 190.6 (180.19)

7. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Deaths
Description: An SAE was defined as any serious adverse event that, at any dose resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or any other situation according to medical or scientific judgment.
Time Frame: From Day 1 up to end of continued access to treatment post-study termination (Day 922)
Population: The analysis was performed on the Safety Population, which included all randomized participants who were exposed to study intervention with the exception of any participants with documented evidence of not having consumed any amount of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Number analyzed (Participants) | 40 | 43 | 42 | 36
Participants
  Serious Adverse Events | 2 | 7 | 2 | 2
  Deaths | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) Leading to Treatment Discontinuation
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Number of participants who discontinued study treatment due to AEs are presented.
Time Frame: From Day 1 up to end of continued access to treatment post-study termination (Day 922)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Number analyzed (Participants) | 40 | 43 | 42 | 36
Participants | 2 | 4 | 5 | 2

9. Secondary Outcome: Number of Participants With AEs Based on Maximum Severity Grades
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. The severity of AEs was defined as per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table) Version 2.1 and was categorized into grades as following: Grade 1 - mild, Grade 2 - moderate, Grade 3 - severe, Grade 4 - Potentially life threatening and Grade 5 - Fatal. Higher grade indicates more severe condition.
Time Frame: From Day 1 up to end of continued access to treatment post-study termination (Day 922)
Population: The analysis was performed on the Safety Population, which included all randomized participants who were exposed to study intervention with the exception of any participants with documented evidence of not having consumed any amount of study intervention. The data presented here is not cumulative data but the number of participants experiencing the adverse event based on maximum grade at the indicated timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Number analyzed (Participants) | 40 | 43 | 42 | 36
Participants
  Grade 1 | 12 | 14 | 17 | 15
  Grade 2 | 19 | 17 | 17 | 10
  Grade 3 | 5 | 5 | 3 | 3
  Grade 4 | 1 | 2 | 1 | 0
  Grade 5 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With AEs of Special Interest (AESI)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Number of participants with AESI (gastrointestinal (GI), nervous system, and psychiatric AEs) are presented.
Time Frame: From Day 1 up to end of continued access to treatment post-study termination (Day 922)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Number analyzed (Participants) | 40 | 43 | 42 | 36
Participants
  AESI (Gastrointestinal) | 15 | 18 | 14 | 14
  AESI (Nervous system) | 7 | 5 | 7 | 3
  AESI (Psychiatric) | 4 | 3 | 4 | 4

11. Secondary Outcome: Number of Participants With Genotypic Resistance
Description: Plasma samples were collected for resistance testing. Genotypic testing was conducted in participants meeting protocol-defined virologic failure (PDVF) criteria. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Only those participants with data available at specified time points have been analyzed.
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: The analysis was performed on the PDVF Population, which included participants with A. virologic non-response (Decrease from Baseline [Day 1] in plasma HIV-1 RNA of ˂1.0 log10 c/mL unless plasma HIV-1 RNA is <200 c/mL by Week 12; confirmed plasma HIV-1 RNA levels ≥200 c/mL at or after Week 24; plasma HIV-1 RNA ≥50 c/mL on repeat testing of Week 24 results and prior to Week 28) and B. virologic rebound (confirmed plasma HIV-1 RNA ≥200 c/mL after confirmed consecutive plasma HIV-1 RNA <50 c/mL).
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Number analyzed (Participants) | 3 | 2 | 5 | 1
Participants
  Baseline (Day 1): number analyzed (Participants) | 3 | 1 | 4 | 1
  Baseline (Day 1) | 0 | 0 | 0 | 0
  Weeks 24: number analyzed (Participants) | 3 | 1 | 4 | 1
  Weeks 24 | 0 | 0 | 0 | 0
  Weeks 48 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Phenotypic Resistance
Description: Plasma samples were collected for resistance testing. Phenotypic testing was conducted in participants meeting PDVF criteria. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and at Weeks 24 and 48
Population: The analysis was performed on the PDVF Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
Number analyzed (Participants) | 3 | 2 | 5 | 1
Participants
  Baseline (Day 1): number analyzed (Participants) | 3 | 1 | 4 | 1
  Baseline (Day 1) | 0 | 0 | 0 | 0
  Weeks 24: number analyzed (Participants) | 3 | 1 | 4 | 1
  Weeks 24 | 0 | 0 | 0 | 0
  Weeks 48 | 0 | 0 | 0 | 0

13. Secondary Outcome: Observed Plasma Concentration at the End of the Dosing Interval (Ctau) of GSK3640254 at Steady State - Week 2
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK3640254. Observed plasma concentration at the end of the dosing interval was determined directly from the concentration-time data.
Time Frame: Pre-dose, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 10, and 24 hours post-dose at Week 2
Population: The analysis was performed on the Intensive PK Population, which included all participants who received at least one dose of GSK3640254, had evaluable drug concentrations reported and where samples were collected according to the intensive PK sampling scheme. Only those participants who received GSK3640254 have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/ milliliter (ng/mL)
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF
Number analyzed (Participants) | 14 | 13 | 18
Nanogram/ milliliter (ng/mL) | 430.5361 (56.5) | 604.8387 (44.2) | 805.2209 (43.7)

14. Secondary Outcome: Observed Plasma Concentration at the End of the Dosing Interval (Ctau) of GSK3640254 at Steady State - Weeks 24 and 48
Description: as for outcome 13
Time Frame: At Weeks 24 and 48
Population: The analysis was performed on the Sparse PK Population, which included all participants who received at least one dose of GSK3640254, had evaluable drug concentrations reported and had samples collected according to the sparse PK sampling scheme. Only those participants who received GSK3640254 and had data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/ milliliter (ng/mL)
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF
Number analyzed (Participants) | 12 | 10 | 13
Nanogram/ milliliter (ng/mL)
  Week 24 | 396.5117 (62.5) | 519.6041 (84.9) | 922.9638 (51.6)
  Week 48: number analyzed (Participants) | 9 | 6 | 6
  Week 48 | 310.9877 (135.4) | 568.0656 (13.4) | 812.4745 (49.1)

15. Secondary Outcome: Area Under the Plasma Drug Concentration-time Curve From Pre-dose to the End of the Dosing Interval (AUC [0-tau]) of GSK3640254 at Steady State
Description: Blood samples were collected at indicated time points for PK analysis of GSK3640254.
Time Frame: Pre-dose, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 10, and 24 hours post-dose at Week 2
Population: The analysis was performed on the Intensive PK Population. Only those participants who received GSK3640254 and had data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/ milliliter (h*ng/mL)
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF
Number analyzed (Participants) | 14 | 13 | 18
Hour*nanogram/ milliliter (h*ng/mL) | 14995.7576 (49.8) | 21212.2480 (44.5) | 30708.2546 (40.1)

16. Secondary Outcome: Maximum Observed Concentration (Cmax) of GSK3640254 at Steady State
Description: Blood samples were collected at indicated time points for PK analysis of GSK3640254.
Time Frame: Pre-dose, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 10, and 24 hours post-dose at Week 2
Population: The analysis was performed on the Intensive PK Population. Only those participants who received GSK3640254 have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF
Number analyzed (Participants) | 15 | 13 | 18
ng/mL | 929.8 (45.9) | 1337.3 (47.7) | 2094.5 (39.2)

17. Secondary Outcome: Observed Pre-dose Plasma Concentration (C0) of GSK3640254 at Steady State
Description: Blood samples were collected at indicated time points for PK analysis of GSK3640254. Observed pre-dose plasma concentration was determined directly from the concentration-time data.
Time Frame: Pre-dose, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 10, and 24 hours post-dose at Week 2
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF
Number analyzed (Participants) | 15 | 13 | 18
ng/mL | 435.9 (54.6) | 603.2 (59.5) | 865.2 (43.4)

18. Secondary Outcome: Time to Cmax (Tmax) of GSK3640254 at Steady State
Description: Blood samples were collected at indicated time points for PK analysis of GSK3640254. Tmax was determined directly from the concentration-time data.
Time Frame: Pre-dose, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 10, and 24 hours post-dose at Week 2
Population: as for outcome 16
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF
Number analyzed (Participants) | 15 | 13 | 18
Hour | 3.0000 [1.900 to 9.017] | 3.4167 [1.000 to 9.000] | 3.4583 [1.917 to 5.000]

19. Secondary Outcome: Steady State Oral Clearance (CLt/F) of GSK3640254
Description: Blood samples were collected at indicated time points for PK analysis of GSK3640254.
Time Frame: Pre-dose, 1, 2, 3, 3.5, 4, 4.5, 5, 6, 10, and 24 hours post-dose at Week 2
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/ hour
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF
Number analyzed (Participants) | 14 | 13 | 18
Liter/ hour | 6.6686 (49.8) | 7.0714 (44.5) | 6.5129 (40.1)

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected from Day 1 up to end of continued access to treatment post-study termination (Day 922).
Description: The study was terminated by the sponsor after primary analysis (at week 48). As prespecified in Statistical analysis plan, AEs were collected up to end of continued access to treatment post-study termination (Day 922).
Arm/Group | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF | GSK3640254 150 mg + ABC/3TC or FTC/TAF | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/43 | 0/42 | 0/36
Serious Adverse Events (participants affected / at risk) | 2/40 | 7/43 | 2/42 | 2/36
Other Adverse Events (participants affected / at risk) | 37/40 | 38/43 | 38/42 | 28/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF (N=40) | GSK3640254 150 mg + ABC/3TC or FTC/TAF (N=43) | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF (N=42) | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF (N=36)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Substance dependence (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3640254 100 mg+ Placebo+ ABC/3TC or FTC/TAF (N=40) | GSK3640254 150 mg + ABC/3TC or FTC/TAF (N=43) | GSK3640254 200 mg+ Placebo+ ABC/3TC or FTC/TAF (N=42) | Dolutegravir (DTG) 50 mg + ABC/3TC or FTC/TAF (N=36)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 7 (8) | 6 (7) | 9 (10)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (8) | 3 (3) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (2)
Pyrexia (General disorders) | 4 (5) | 4 (4) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 10 (12) | 12 (12) | 6 (7) | 10 (13)
Chlamydial infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Gonorrhoea (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 4 (4) | 3 (3) | 4 (5)
Monkeypox (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (5) | 3 (4) | 3 (5) | 3 (6)
Pharyngitis (Infections and infestations) | 4 (4) | 4 (5) | 1 (1) | 3 (3)
Respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 3 (3) | 1 (1) | 3 (3) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 3 (3) | 3 (5) | 1 (1)
Urethritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 4 (4) | 7 (10) | 3 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 2 (2) | 3 (4)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT04493216/Prot_002.pdf
  • Statistical Analysis Plan (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT04493216/SAP_004.pdf